CLINICAL TRIAL: NCT04692857
Title: Ultrasound-guided Fascia Iliaca Compartment Block After Hip Fracture : the Effect of the Local Anesthetic Volume on the Quality of Preoperative Analgesia
Brief Title: US-guided FICB After Hip Fracture: the Effect of the Local Anesthetic Volume on the Quality of Preoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mechaal Benali, professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTEM VOL FIBSI
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 30 (Experimental): participants received a supra inguinal fascia iliaca compartment block with 30 ml of 0.2% ropivacaine
  Interventions: Procedure: supra inguinal fascia iliaca block
- group 40 (Experimental): participants received a supra inguinal fascia iliaca compartment block with 40 ml of 0.2% ropivacaine
  Interventions: Procedure: supra inguinal fascia iliaca block
- group 50 (Experimental): participants received a supra inguinal fascia iliaca compartment block with 50 ml of 0.2% ropivacaine
  Interventions: Procedure: supra inguinal fascia iliaca block

INTERVENTIONS:
Procedure: supra inguinal fascia iliaca block — injection of 30,40 or 50 ml of 0.2 ropivacaine .

SUMMARY:
participants were randomly divided into three groups : group 30 , group 40 and group 50 . for all the three groups an ultrasound guided supra-inguinal fascia iliaca block had been performed.

for group 30 ,a volume of 30 ml of 0,2 % ropivacaine had been injected for group 40 ,a volume of 40 ml of 0,2 % ropivacaine had been injected for group 50 ,a volume of 50 ml of 0,2 % ropivacaine had been injected

DETAILED DESCRIPTION:
participants were randomly divided into three groups : group 30 , group 40 and group 50 . for all the three groups an ultrasound guided supra-inguinal fascia iliaca block had been performed.

A linear ultrasound probe was placed in the sagittal plane to obtain an image of the superior iliac spine.the fascia iliaca and sartorious,iliopsoas,and oblique internal muscles were identified by sliding the probe medially. After identifiying the "bow-tie sign"formed by the muscle fascias , an 50 mm needle was introduced 1-2 cm inferior to the inguinal ligament.using an in-plane approch, the fascia iliaca was penetrated and hydrodissected , separating the fascia iliaca from the iliac muscle. in this created space a total volume of 30 ml, 40ml or 50ml of 0.2% ropivacaine was injected , respectively to group 30 ,group 40 and group 50 .

pain score at rest and with a straight leg raise of the affected limb to 15 degrees were assessed before and 30 minutes after block performance.

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 65 years , american society of anesthesiologists physical status I to III , and with body mass index (BMI) of 35 kg/m² or less , undergoing hip fracture surgical repair .

Exclusion Criteria:

* inability or refusal to sign informed consent
* younger than 65 years
* BMI greater than 35 kg/m²
* presence of contraindications for regional nerve block or spinal anesthesia
* impaired cognition or dementia
* multiple fractures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
change in pain score on movement | before and 30 minutes after block placement
  change in verbal ranking scale(( vrs) with 0 indicating no pain and 10 indicating the worst imaginable pain)) during passive leg elevation to 15 degrees of the affected limb , before and 30 minutes after block placement

SECONDARY OUTCOMES:
change in pain score at rest | before and 30 minutes after block placement
  change in verbal ranking scale(( vrs) with 0 indicating no pain and 10 indicating the worst imaginable pain)) at rest, before and 30 minutes after block placement
assessement of sensory block | 30 minutes after block placement
  sensory assessment of Femoral nerve , obturator nerve, and lateral femoral cutaneous nerve using the cold test . in the anterior , medial and lateral aspects of the thigh.

CONTACTS AND LOCATIONS:
Overall Officials: mechaal benali, PROFESSOR, Study Chair — university manar Tunis tunisia
Locations (1):
- Mechaal Benali, Nabeul, Mrezga, Tunisia

IPD SHARING:
Plan to Share IPD: No